CLINICAL TRIAL: NCT06048471
Title: High Tone Therapy for Chemotherapy Induced Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Hospital Association (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HiTop Protocol v.1.3
Record Dates: First submitted 2020-03-02; First posted 2023-09-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Electrical Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HiTop (Experimental)
  Interventions: Other: HiTop
- Sham stimulation (Sham Comparator)
  Interventions: Other: HiTop

INTERVENTIONS:
Other: HiTop — High tone transcutaneous electrical stimulation

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN), a side effect of antineoplastic medication, was reported to occur in about 68% of the patients receiving chemotherapy. CIPN does not only limit quality of life due to neuropathic symptoms but also may lead to dose reductions or premature interruption of therapy and thus to suboptimal cancer treatment.

Patients with neuropathy suffer from sensory disturbances as tingling, numbness, burning pain or sleep disturbances and even though numerous drugs are available, it is still difficult to sufficiently control these Symptoms.

High tone therapy / high tone external muscle stimulation (HTEMS) seems to be an effective treatment for neuropathic symptoms. Previous studies observed promising results in diabetics and chronic kidney disease (CKD) patients.

To date, there is no investigation on HTEMS in patients with chemotherapy induced neuropathy.

Therefore, this aim of this project is to test if HTEMS would bring about a stronger decrease in neuropathic symptoms in this specific patient group, compared to a placebo treatment.

The primary objective is the alleviation of paresthesias. The secondary objective focuses on detailed symptoms of neuropathiy as well as on health-related quality of life.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically verified colorectal cancer and adjuvant treatment with a platin derivate (e.g., cisplatin, oxaliplatin): This group was chosen due to relatively high risk of neuropathy due to this special therapeutic agent 1,9.
* Cumulative dose of at least 3 cycles
* Interval of 2 weeks since the last chemotherapeutic cycle in order to prevent false worsenings due to delayed neurotoxic effects
* Life expectancy of at least 3 months
* Stable medication (no changes of especially pain medication during the study)
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2 (that is, the capability to walk and to spend less than 50% of waking hours sitting or lying)
* Ability to walk (with or without aids)
* European Organisation for Research and Treatment of Cancer (EORTC) common toxicity criteria (CTC) peripheral sensory neuropathy grade 1 or 2
* Intensity of paresthesias of 3/10 or higher on the Numeric Rating Scale (NRS)

Exclusion criteria:

* Prevalent neuropathy of different etiology
* Serious central-neurological or psychiatric disorder that would interfer with a proper order of the study, according to the judgement of the investigators
* Epilepsy
* Minors or persons unable to give informed consent
* Current neurotoxic medication
* Implanted pacemakers or defibrillators
* Pregnancy
* Wounds in the area to be treated, acute local or systemic infection
* Peripheral arterial occlusive disease > grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Intensity of paresthesia | 5 weeks
  NRS scale

SECONDARY OUTCOMES:
health related Quality of life (QOL), detailed symptroms of neuropathy | 5 weeks
  EORTC C30, CIPN 20, Neuropathy symptom scale (NSS), NRS scales

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Donaustadt, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wakolbinger-Habel R, Reinweber M, Alakraa M, Riener I, Scheffold BE, Racz K, Selimi F, Straub C, Jauker J, Bily W, Niedersuss-Beke D, Mayrhofer K, Paternostro-Sluga T. Home-based high tone therapy may alleviate chemotherapy-induced neuropathic symptoms in patients with colorectal cancer: A randomized double-blind placebo-controlled pilot evaluation. Support Care Cancer. 2024 Jan 27;32(2):134. doi: 10.1007/s00520-024-08331-7. PMID 38280118

DOCUMENTS (1):
  • Study Protocol (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06048471/Prot_000.pdf